CLINICAL TRIAL: NCT04505020
Title: The Innovation of 3D Printing for Preoperative Planning in Hip Preservation Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ivan Wong, MD, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3DPRINT
Record Dates: First submitted 2020-04-30; First posted 2020-08-07 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Femoro Acetabular Impingement
Keywords: Femoroacetabular Impingement; Cam lesion; 3D printing; Pre-operative planning
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Intervention Model Description: Patients that have consented to the study will be randomized into four groups with a 50% chance of being in either group. The two treatment groups are 1) conventional preoperative imaging (X-ray, CT, and MRI) only 2) those that have had a 3D printed model created in addition to conventional imaging. There will be 40 patients in each group. Randomization will be done with a computer random number generator. Both groups will undergo routine pre-operative imaging but one group will also have a 3D print made from the 3D CT reconstruction. Both patient groups will undergo hip arthroscopy for treatment of their FAI.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded/masked to the treatment (if they do or don't receive a 3D printed model of their hip) they receive until the end of the study. Patients will still be aware of the details of their surgical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D Print + Conventional imaging (Experimental): Patients in this group allocation will receive a 3D reconstruction of their hip in addition to conventional preoperative imaging (X-ray, CT, and MRI) only for the use of pre-operative and intra-operative planning for their hip arthroscopy (FAI) procedure.
  Interventions: Other: 3D Print + Conventional imaging
- Conventional Imaging (Other): Patients in this group allocation will receive conventional preoperative imaging (X-ray, CT, and MRI) only for the use of pre-operative and intra-operative planning for their hip arthroscopy (FAI) procedure.
  Interventions: Other: Conventional imaging

INTERVENTIONS:
Other: 3D Print + Conventional imaging — This group will have a 3D reconstruction of their hip printed using a 3D printer so that the PI can use it in their pre and intra-operative planning along with traditional imaging.
  Arms: 3D Print + Conventional imaging
Other: Conventional imaging — This group will have CT, MRI and X-Ray imaging completed so that the PI can use it in their pre and intra-operative planning.
  Arms: Conventional Imaging

SUMMARY:
This is a randomized controlled trial (RCT) to evaluate the introduction of a 3D printed model into the pre and intra-operative planning for arthroscopic femoroacetabular impingement (FAI) surgery. The RCT will look to place patients into one of two treatment groups: 1) conventional preoperative imaging (X-ray, CT, and MRI) only and 2) those that have had a 3D printed model created in addition to the conventional imaging.

DETAILED DESCRIPTION:
In this study, we investigate the use of 3D models during pre and intra-operative planning could improve the success of hip arthroscopy and reduce the incidence of revision cases. By adding an adjunct to the common suite of pre-operative imaging modalities (X-ray, MRI and CT), we can change the surgeon's understanding of each patient's individual morphology with a tactile physical model. This study will compare the success of hip arthroscopy in patients with or without 3D printed models (in addition to traditional pre-operative imaging).

This will be a single-center, blinded observer, randomized controlled trial of 80 patients performed at the Halifax Infirmary, Queen Elizabeth II Health Sciences Center in Halifax, Nova Scotia. Patients with cam-type FAI involved in the study will be approached by the surgeon, Dr. Ivan Wong, or a delegate regarding the study during a pre-operative visit. Following a detailed discussion of the risks/benefits/alternatives of this study, the patient will be provided with a copy of the informed consent to review, if they demonstrate an interest in the study. If the patient wishes to be enrolled in the study, the research team will obtain patient consent for the study according to the Division of Orthopaedic Surgery and Nova Scotia Health Authority (NSHA) institutional protocols.

In the pre-operative period, there will be no additional time requirements for the participant, except for the informed consent process for the study. Routine X-ray radiographs, as well as a pre-operative MRI and CT scan, will be obtained for all subjects undergoing FAI surgery. The participants will not be exposed to any additional radiation. Subjects will complete a structured clinical examination conducted by a sports medicine fellowship-trained orthopaedic consultant. The patient will also complete pre-operative questionnaires.

Patients that have consented to the study will be randomized into two groups with a 50% chance of being in either group. Randomization will be done with a computer random number generator. Both groups will undergo routine pre-operative imaging but one group will also have a 3D print made from the 3D CT reconstruction. All patient groups will undergo hip arthroscopy for the treatment of their FAI.

ELIGIBILITY:
Inclusion Criteria:

* Radiological proven diagnosis of cam-type femoroacetabular impingement (FAI)

Exclusion Criteria:

* Patients with advanced arthritis (Tonnis Grade III or Kellgren-Lawrence Grade III or IV or evidence of less than 2 mm of joint space, as determined by conventional radiographs.)
* Patients with 1cm2 (or greater) of cartilage delamination in the hip
* Patients with type III or IV heterotopic ossification
* Patients with avascular necrosis
* Patients who are unable to provide informed consent
* Patients who are undergoing revision hip arthroscopy
* Patients who are pregnant
* Patients who have the presence of local or systemic infection
* Patients with an inability to cooperate with and/or comprehend post-operative instructions
* Patients with nonvascular surgical sites (MRI proven)
* Patients with cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Measure of CAM resection | Change in Pre-op measurements compared to 2 weeks post-operatively
  Our primary outcome for this study is the resection of cam impingement according to alpha-angle on post-operative anterior-posterior (AP) and frog leg X-ray views.
Measure of CAM resection | Change in Pre-op measurements compared to 6 months post-operatively
  Our primary outcome for this study is the resection of cam impingement according to alpha-angle on post-operative anterior-posterior (AP) and frog leg X-ray views.
Measure of CAM resection | Change in Pre-op measurements compared to 24 months post-operatively
  Our primary outcome for this study is the resection of cam impingement according to alpha-angle on post-operative anterior-posterior (AP) and frog leg X-ray views.

SECONDARY OUTCOMES:
Differences in post-operative patient reported outcomes: iHOT-33 | Change in outcomes 24 months post operatively compared to Pre-operatively
  The secondary outcome is the differences in post-operative patient reported outcomes for the international hip outcome tool (iHOT-33) when compared to a pre-operative baseline. (Scores for the International hip outcome tool range from 0-100 where higher values represent better outcomes)
Differences in post-operative patient reported outcomes: NAHS | Change in outcomes 24 months post operatively compared to Pre-operatively
  The secondary outcome is the differences in post-operative patient reported outcomes for the Non-arthritic Hip Score (NAHS) when compared to a pre-operative baseline. (Scores for the Non-arthritic Hip Score range from 0-80 where higher values represent better outcomes).
Differences in post-operative patient reported outcomes: EQ5D | Change in outcomes 24 months post operatively compared to Pre-operatively
  The secondary outcome is the differences in post-operative patient reported outcomes for the European Quality of Life Questionnaire (EQ-5D) when compared to a pre-operative baseline. (Scores for EQ-5D range from 1-5 in 5 categories where lower values represent better outcomes in each category).
Differences in post-operative patient reported outcomes: EQ5D-VAS | Change in outcomes 24 months post operatively compared to Pre-operatively
  The secondary outcome is the differences in post-operative patient reported outcomes for the European Quality of Life Questionnaire-Visual Analog Scale (EQ-5D-VAS) when compared to a pre-operative baseline. (Scores for EQ-5D-VAS range from 0-100 where higher values represent better outcomes).
Differences in post-operative patient reported outcomes: VR-12 | Change in outcomes 24 months post operatively compared to Pre-operatively
  The secondary outcome is the differences in post-operative patient reported outcomes for the Veteran's RAND 12 Item Health Survey (VR-12) when compared to a pre-operative baseline. (Scores for VR-12 range from 0-100 where higher values represent better outcomes).
Differences in post-operative patient reported outcomes: HOS-Usual Activities | Change in outcomes 24 months post operatively compared to Pre-operatively
  The secondary outcome is the differences in post-operative patient reported outcomes for the Hip Outcome Score for usual activities (HOS-UA) when compared to a pre-operative baseline. (Scores for HOS range from 0-68 where higher values represent better outcomes).
Differences in post-operative patient reported outcomes: HOS-Sport | Change in outcomes 24 months post operatively compared to Pre-operatively
  The secondary outcome is the differences in post-operative patient reported outcomes for the Hip Outcome Score for sports (HOS-S) when compared to a pre-operative baseline. (Scores for HOS range from 0-30 where higher values represent better outcomes).

OTHER OUTCOMES:
The number of times conventional imaging and 3D prints are referenced intra-operatively. | During surgery only
  Another secondary outcome is the number of times each of the following are referenced intra-operatively: X-Rays, MRI, MRA, CT, CT with 3D reconstruction and 3D model of patient's hip. Additionally the number of X-Ray images taken intra-operatively will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wong, Dr., Principal Investigator — Nova Scotia Health Authority
Locations (1):
- 5955 Veterans' Memorial Lane Room 2106, VMB, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.